CLINICAL TRIAL: NCT00397943
Title: Safety, Reactogenicity & Immunogenicity of 2 Formulations of Tuberculosis Vaccine GSK692342 Administered Intramuscularly According to a Schedule of 0, 1 Month, to Healthy Adults Aged 18 to 50 Years
Brief Title: Safety and Immunogenicity of 2 Formulations of Tuberculosis Vaccine GSK692342 Given at 0,1 Months to Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 106227; 106228 (Other: GSK); 108736 (Other: GSK); 108738 (Other: GSK); 2005-004497-24 (EudraCT Number)
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Tuberculosis
Keywords: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- M72/AS01B Group (Experimental): Healthy male or female subjects, between and including 18 to 50 years of age, who received 2 doses of M72/AS01B vaccine, administered intramuscularly in the deltoid muscle of the non-dominant arm at Month 0 and Month 1.
  Interventions: Biological: GSK's candidate Mycobacterium tuberculosis vaccine 692342
- M72/AS02A Group (Experimental): Healthy male or female subjects, between and including 18 to 50 years of age, who received 2 doses of M72/AS02A vaccine, administered intramuscularly in the deltoid muscle of the non-dominant arm at Month 0 and Month 1.
  Interventions: Biological: GSK's candidate Mycobacterium tuberculosis vaccine 692342
- Mtb72F/AS02A Group (Active Comparator): Healthy male or female subjects, between and including 18 to 50 years of age, who received 2 doses of the comparator Mtb72F/AS02A vaccine, administered intramuscularly in the deltoid muscle of the non-dominant arm at Month 0 and Month 1.
  Interventions: Biological: Comparator vaccine with recombinant Mycobacterium tuberculosis antigen and adjuvant system
- Non-adjuvanted Group (Active Comparator): Healthy male or female subjects, between and including 18 to 50 years of age, who received 2 doses of the comparator GSK Biologicals' candidate recombinant M. tuberculosis vaccine, non-adjuvanted, administered intramuscularly in the deltoid muscle of the non-dominant arm at Month 0 and Month 1.
  Interventions: Biological: Comparator vaccine with recombinant Mycobacterium tuberculosis antigen and physiological saline
- Control Group (Placebo Comparator): Healthy male or female subjects, between and including 18 to 50 years of age, who received 2 doses of the adjuvant system alone, administered intramuscularly in the deltoid muscle of the non-dominant arm at Month 0 and Month 1.
  Interventions: Biological: Control vaccine with the adjuvant system.

INTERVENTIONS:
Biological: GSK's candidate Mycobacterium tuberculosis vaccine 692342 — Intramuscular injection, 2 doses at 0, 1 month
  Arms: M72/AS01B Group; M72/AS02A Group
Biological: Comparator vaccine with recombinant Mycobacterium tuberculosis antigen and adjuvant system — Intramuscular injection, 2 doses at 0, 1 month
  Arms: Mtb72F/AS02A Group
Biological: Comparator vaccine with recombinant Mycobacterium tuberculosis antigen and physiological saline — Intramuscular injection, 2 doses at 0, 1 month
  Arms: Non-adjuvanted Group
Biological: Control vaccine with the adjuvant system. — Intramuscular injection, 2 doses at 0, 1 month
  Arms: Control Group

SUMMARY:
This study will assess the safety and immunogenicity of 2 different formulations of tuberculosis vaccine GSK692342 in healthy adults.

DETAILED DESCRIPTION:
The study is designed to have a vaccination phase (includes screening, 2 doses of vaccine 1 month apart and follow-up until 1 month post dose 2), which will be performed in an observer blinded manner. This will be followed by 3 years of follow-up which will continue in an open manner.

No new subjects will be recruited at the follow-up phase. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol
* A male or female between, and including, 18 and 50 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject prior to any study procedure.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Subjects must have PPD negative skin reactivity (0 mm induration 48 to 72 hours after PPD skin test administration).
* Clinically normal laboratory values for creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST), complete blood count (CBC) and differential, haemoglobin, platelet count and urinalysis.
* Seronegative for human immunodeficiency virus-1 and 2 (HIV 1/2) antibodies, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibodies
* If the subject is female, she must be of non-childbearing potential, or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.
* No evidence of pulmonary pathology (i.e. acute or chronic pulmonary disease; past TB infection/disease) as confirmed by chest X-ray.

Exclusion Criteria:

* History of previous exposure to experimental products containing components of the experimental vaccine.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose.
* Any chronic drug therapy to be continued during the study period. Vitamins and/or dietary supplements, herbal medications, birth control pills, anti-histamines for seasonal allergies, SSRIs (e.g. Prozac, Zoloft, Paxil), NSAIDs (nonsteroidal anti-inflammatory drugs e.g. aspirin, ibuprofen), and acetaminophen are allowed.
* History of documented exposure to Mycobacterium tuberculosis.
* History of prior vaccination with experimental Mycobacterium tuberculosis vaccines.
* Administration of any immunoglobulins, any immunotherapy and/or any blood products within the 3 months preceding the first dose of study vaccination, or planned administrations during the study period.
* Participation in another experimental protocol during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition; or family history of congenital or hereditary immunodeficiency.
* History of hypersensitivity to vaccines or vaccine components
* History of any acute or chronic illness or medication that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.
* Volunteers with a personal history of autoimmune disease or who describe a first-degree relative with clearly documented autoimmune disease.
* History of any neurological disorders or seizures.
* History of chronic alcohol consumption and/or drug abuse.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects.
* Pregnant female, lactating female or female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2006-11-15 (Actual); Primary Completion 2009-12-01 (Actual); Study Completion 2009-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Leroux-Roels I, Forgus S, De Boever F, Clement F, Demoitie MA, Mettens P, Moris P, Ledent E, Leroux-Roels G, Ofori-Anyinam O; M72 Study Group. Improved CD4(+) T cell responses to Mycobacterium tuberculosis in PPD-negative adults by M72/AS01 as compared to the M72/AS02 and Mtb72F/AS02 tuberculosis candidate vaccine formulations: a randomized trial. Vaccine. 2013 Apr 19;31(17):2196-206. doi: 10.1016/j.vaccine.2012.05.035. Epub 2012 May 27. PMID 22643213
- [Derived] Moris P, Bellanger A, Ofori-Anyinam O, Jongert E, Yarzabal Rodriguez JP, Janssens M. Whole blood can be used as an alternative to isolated peripheral blood mononuclear cells to measure in vitro specific T-cell responses in human samples. J Immunol Methods. 2021 May;492:112940. doi: 10.1016/j.jim.2020.112940. Epub 2021 Jan 23. PMID 33493551

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Started | 40 | 40 | 10 | 10 | 10
Completed | 28 | 31 | 10 | 10 | 10
Not Completed | 12 | 9 | 0 | 0 | 0
Not completed — Unspecified reasons | 12 | 9 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group | Total
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.0 (6.50) | 26.4 (7.97) | 28.5 (6.95) | 24.8 (5.33) | 25.9 (7.95) | 25.89 (7.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 9 | 4 | 7 | 67
  Male | 16 | 17 | 1 | 6 | 3 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-Arabic/North African heritage | 0 | 1 | 0 | 0 | 0 | 1
  White-Caucasian/European heritage | 38 | 39 | 10 | 10 | 10 | 107
  Unspecified | 2 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) follow-up period after each vaccine dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
Participants
  Any Pain, Dose 1 | 38 | 40 | 9 | 1 | 10
  Grade 3 Pain, Dose 1 | 7 | 5 | 4 | 0 | 1
  Any Redness, Dose 1 | 4 | 2 | 0 | 0 | 1
  Grade 3 Redness, Dose 1 | 2 | 2 | 0 | 0 | 0
  Any Swelling, Dose 1 | 4 | 8 | 2 | 0 | 2
  Grade 3 Swelling, Dose 1 | 2 | 3 | 0 | 0 | 1
  Any Pain, Dose 2 | 39 | 37 | 9 | 2 | 10
  Grade 3 Pain, Dose 2 | 7 | 4 | 2 | 0 | 0
  Any Redness, Dose 2 | 10 | 2 | 1 | 1 | 1
  Grade 3 Redness, Dose 2 | 6 | 0 | 0 | 1 | 1
  Any Swelling, Dose 2 | 7 | 9 | 4 | 1 | 2
  Grade 3 Swelling, Dose 2 | 1 | 3 | 2 | 1 | 1
  Any Pain, Across doses | 40 | 40 | 10 | 2 | 10
  Grade 3 Pain, Across doses | 13 | 6 | 4 | 0 | 1
  Any Redness, Across doses | 12 | 4 | 1 | 1 | 2
  Grade 3 Redness, Across doses | 6 | 2 | 0 | 1 | 1
  Any Swelling, Across doses | 9 | 10 | 5 | 1 | 3
  Grade 3 Swelling, Across doses | 3 | 4 | 2 | 1 | 1

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], gastrointestinal symptoms and headache. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 7-day (Days 0-6) follow-up period after each vaccine dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
Participants
  Any Fatigue, Dose 1 | 27 | 21 | 6 | 2 | 3
  Grade 3 Fatigue, Dose 1 | 0 | 1 | 0 | 1 | 0
  Related Fatigue, Dose 1 | 26 | 19 | 5 | 2 | 3
  Any Fever, Dose 1 | 5 | 2 | 1 | 0 | 1
  Grade 3 Fever, Dose 1 | 0 | 0 | 0 | 0 | 0
  Related Fever, Dose 1 | 3 | 2 | 0 | 0 | 1
  Any Gastrointestinal symptoms, Dose 1 | 9 | 7 | 3 | 2 | 1
  Grade 3 Gastrointestinal symptoms, Dose 1 | 1 | 0 | 0 | 0 | 0
  Related Gastrointestinal symptoms, Dose 1 | 6 | 7 | 1 | 1 | 1
  Any Headache, Dose 1 | 19 | 12 | 9 | 2 | 3
  Grade 3 Headache, Dose 1 | 0 | 0 | 1 | 0 | 0
  Related Headache, Dose 1 | 15 | 11 | 4 | 1 | 3
  Any Fatigue, Dose 2 | 33 | 24 | 7 | 2 | 6
  Grade 3 Fatigue, Dose 2 | 4 | 2 | 0 | 0 | 1
  Related Fatigue, Dose 2 | 33 | 23 | 7 | 1 | 4
  Any Fever, Dose 2 | 24 | 10 | 4 | 0 | 1
  Grade 3 Fever, Dose 2 | 0 | 0 | 0 | 0 | 1
  Related Fever, Dose 2 | 24 | 10 | 4 | 0 | 0
  Any Gastrointestinal symptoms, Dose 2 | 18 | 10 | 3 | 2 | 2
  Grade 3 Gastrointestinal symptoms, Dose 2 | 2 | 2 | 0 | 1 | 0
  Related Gastrointestinal symptoms, Dose 2 | 17 | 8 | 3 | 1 | 1
  Any Headache, Dose 2 | 32 | 22 | 6 | 2 | 4
  Grade 3 Headache, Dose 2 | 8 | 2 | 0 | 0 | 1
  Related Headache, Dose 2 | 32 | 19 | 6 | 1 | 3
  Any Fatigue, Across doses | 36 | 29 | 8 | 3 | 6
  Grade 3 Fatigue, Across doses | 4 | 3 | 0 | 1 | 1
  Related Fatigue, Across doses | 36 | 28 | 7 | 3 | 5
  Any Fever, Across doses | 25 | 10 | 4 | 0 | 1
  Grade 3 Fever, Across doses | 0 | 0 | 0 | 0 | 1
  Related Fever, Across doses | 25 | 10 | 4 | 0 | 1
  Any Gastrointestinal symptoms, Across doses | 23 | 10 | 5 | 2 | 2
  Grade 3 Gastrointestinal symptoms, Across doses | 3 | 2 | 0 | 1 | 0
  Related Gastrointestinal symptoms, Across doses | 20 | 9 | 4 | 2 | 2
  Any Headache, Across doses | 33 | 27 | 9 | 3 | 5
  Grade 3 Headache, Across doses | 8 | 2 | 1 | 0 | 1
  Related Headache, Across doses | 32 | 24 | 7 | 2 | 5

3. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (Days 0-29) follow-up period after each vaccine dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
Participants
  Any AE(s) | 37 | 33 | 10 | 7 | 7
  Grade 3 AE(s) | 12 | 7 | 4 | 2 | 1
  Related AE(s) | 31 | 21 | 8 | 2 | 4

4. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the Active Vaccination Phase (from Day 0 up to Month 2)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
Participants | 0 | 0 | 1 | 0 | 0

5. Primary Outcome: Number of Subjects With SAEs
Description: as for outcome 4
Time Frame: From Month 2 up to Month 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
Participants | 2 | 0 | 0 | 0 | 1

6. Primary Outcome: Number of Subjects With SAEs
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Note: Follow-up during Year 2 continued only for the M72/AS01B Group and M72/AS02A Group.
Time Frame: From Month 12 up to Month 24
Population: The analysis was performed on the Total Vaccinated cohort (all subjects with at least one vaccine administration documented and with the symptom sheet filled in) and focused on the subjects included in the Year 2 Safety Follow-Up (M72/AS01B and M72/AS02A groups).
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01B Group | M72/AS02A Group
Number analyzed (Participants) | 32 | 37
Participants | 0 | 0

7. Primary Outcome: Number of Subjects With SAEs
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Note: Follow-up during Year 3 continued only for the M72/AS01B Group and M72/AS02A Group.
Time Frame: From Month 24 up to Month 36
Population: The analysis was performed on the Total Vaccinated cohort (all subjects with at least one vaccine administration documented and with the symptom sheet filled in) and focused on the subjects included in the Year 3 Safety Follow-Up (M72/AS01B and M72/AS02A groups).
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01B Group | M72/AS02A Group
Number analyzed (Participants) | 28 | 31
Participants | 0 | 0

8. Primary Outcome: Number of Subjects With Normal or Abnormal Haematological and Biochemical Levels
Description: Among haematological and biochemical parameters assessed were Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Basophils, Creatinine, Eosinophils, Haemoglobin, Haematocrite, Lymphocytes, Monocytes, Neutrophils, Platelets, Red blood cells (RBC), White blood cells (WBC). Inside = within laboratory reference range; Above = above laboratory reference range; Below = below laboratory reference range.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
Participants
  ALT, Inside | 39 | 39 | 9 | 10 | 10
  ALT, Above | 0 | 1 | 1 | 0 | 0
  ALT, Below | 1 | 0 | 0 | 0 | 0
  ALT, Missing | 0 | 0 | 0 | 0 | 0
  AST, Inside | 39 | 40 | 10 | 10 | 10
  AST, Above | 1 | 0 | 0 | 0 | 0
  AST, Below | 0 | 0 | 0 | 0 | 0
  AST, Missing | 0 | 0 | 0 | 0 | 0
  Basophils, Inside | 40 | 40 | 10 | 10 | 10
  Basophils, Above | 0 | 0 | 0 | 0 | 0
  Basophils, Below | 0 | 0 | 0 | 0 | 0
  Basophils, Missing | 0 | 0 | 0 | 0 | 0
  Creatinine, Inside | 39 | 39 | 9 | 10 | 10
  Creatinine, Above | 1 | 0 | 0 | 0 | 0
  Creatinine, Below | 0 | 1 | 1 | 0 | 0
  Creatinine, Missing | 0 | 0 | 0 | 0 | 0
  Eosinophils, Inside | 37 | 40 | 10 | 10 | 10
  Eosinophils, Above | 3 | 0 | 0 | 0 | 0
  Eosinophils, Below | 0 | 0 | 0 | 0 | 0
  Eosinophils, Missing | 0 | 0 | 0 | 0 | 0
  Haemoglobin, Inside | 40 | 38 | 10 | 9 | 10
  Haemoglobin, Above | 0 | 1 | 0 | 0 | 0
  Haemoglobin, Below | 0 | 1 | 0 | 1 | 0
  Haemoglobin, Missing | 0 | 0 | 0 | 0 | 0
  Haematocrite, Inside | 37 | 37 | 10 | 9 | 10
  Haematocrite, Above | 0 | 0 | 0 | 0 | 0
  Haematocrite, Below | 3 | 3 | 0 | 1 | 0
  Haematocrite, Missing | 0 | 0 | 0 | 0 | 0
  Lymphocytes, Inside | 39 | 39 | 10 | 8 | 8
  Lymphocytes, Above | 0 | 0 | 0 | 1 | 1
  Lymphocytes, Below | 1 | 1 | 0 | 1 | 1
  Lymphocytes, Missing | 0 | 0 | 0 | 0 | 0
  Monocytes, Inside | 29 | 32 | 8 | 6 | 6
  Monocytes, Above | 10 | 8 | 1 | 4 | 4
  Monocytes, Below | 1 | 0 | 1 | 0 | 0
  Monocytes, Missing | 0 | 0 | 0 | 0 | 0
  Neutrophils, Inside | 38 | 38 | 9 | 9 | 9
  Neutrophils, Above | 1 | 1 | 1 | 0 | 0
  Neutrophils, Below | 1 | 1 | 0 | 1 | 1
  Neutrophils, Missing | 0 | 0 | 0 | 0 | 0
  Platelets, Inside | 38 | 39 | 10 | 9 | 10
  Platelets, Above | 0 | 0 | 0 | 1 | 0
  Platelets, Below | 2 | 1 | 0 | 1 | 0
  Platelets, Missing | 0 | 0 | 0 | 0 | 0
  RBC, Inside | 40 | 39 | 10 | 10 | 10
  RBC, Above | 0 | 0 | 0 | 0 | 0
  RBC, Below | 0 | 1 | 0 | 0 | 0
  RBC, Missing | 0 | 0 | 0 | 0 | 0
  WBC, Inside | 36 | 36 | 10 | 9 | 9
  WBC, Above | 3 | 2 | 0 | 0 | 0
  WBC, Below | 1 | 2 | 0 | 1 | 1
  WBC, Missing | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Subjects With Normal and Abnormal Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: At Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
Participants
  ALT, Inside | 38 | 40 | 10 | 10 | 10
  ALT, Above | 2 | 0 | 0 | 0 | 0
  ALT, Below | 0 | 0 | 0 | 0 | 0
  ALT, Missing | 0 | 0 | 0 | 0 | 0
  AST, Inside | 39 | 39 | 10 | 10 | 10
  AST, Above | 1 | 1 | 0 | 0 | 0
  AST, Below | 0 | 0 | 0 | 0 | 0
  AST, Missing | 0 | 0 | 0 | 0 | 0
  Basophils, Inside | 40 | 40 | 10 | 10 | 10
  Basophils, Above | 0 | 0 | 0 | 0 | 0
  Basophils, Below | 0 | 0 | 0 | 0 | 0
  Basophils, Missing | 0 | 0 | 0 | 0 | 0
  Creatinine, Inside | 37 | 39 | 10 | 10 | 9
  Creatinine, Above | 2 | 0 | 0 | 0 | 1
  Creatinine, Below | 1 | 1 | 0 | 0 | 0
  Creatinine, Missing | 0 | 0 | 0 | 0 | 0
  Eosinophils, Inside | 39 | 39 | 10 | 10 | 10
  Eosinophils, Above | 1 | 1 | 0 | 0 | 0
  Eosinophils, Below | 0 | 0 | 0 | 0 | 0
  Eosinophils, Missing | 0 | 0 | 0 | 0 | 0
  Haemoglobin, Inside | 40 | 38 | 10 | 9 | 10
  Haemoglobin, Above | 0 | 0 | 0 | 0 | 0
  Haemoglobin, Below | 0 | 2 | 0 | 1 | 0
  Haemoglobin, Missing | 0 | 0 | 0 | 0 | 0
  Haematocrite, Inside | 39 | 36 | 10 | 9 | 10
  Haematocrite, Above | 0 | 0 | 0 | 0 | 0
  Haematocrite, Below | 1 | 4 | 0 | 1 | 0
  Haematocrite, Missing | 0 | 0 | 0 | 0 | 0
  Lymphocytes, Inside | 40 | 38 | 8 | 10 | 8
  Lymphocytes, Above | 0 | 1 | 1 | 0 | 1
  Lymphocytes, Below | 0 | 1 | 1 | 0 | 1
  Lymphocytes, Missing | 0 | 0 | 0 | 0 | 0
  Monocytes, Inside | 29 | 33 | 7 | 9 | 8
  Monocytes, Above | 11 | 7 | 3 | 1 | 2
  Monocytes, Below | 0 | 0 | 0 | 0 | 0
  Monocytes, Missing | 0 | 0 | 0 | 0 | 0
  Neutrophils, Inside | 40 | 39 | 7 | 10 | 8
  Neutrophils, Above | 0 | 1 | 1 | 0 | 1
  Neutrophils, Below | 0 | 0 | 2 | 0 | 1
  Neutrophils, Missing | 0 | 0 | 0 | 0 | 0
  Platelets, Inside | 40 | 39 | 10 | 9 | 10
  Platelets, Above | 0 | 0 | 0 | 0 | 0
  Platelets, Below | 0 | 1 | 0 | 1 | 0
  Platelets, Missing | 0 | 0 | 0 | 0 | 0
  RBC, Inside | 40 | 39 | 10 | 10 | 10
  RBC, Above | 0 | 0 | 0 | 0 | 0
  RBC, Below | 0 | 1 | 0 | 0 | 0
  RBC, Missing | 0 | 0 | 0 | 0 | 0
  WBC, Inside | 37 | 38 | 9 | 10 | 10
  WBC, Above | 2 | 0 | 0 | 0 | 0
  WBC, Below | 1 | 2 | 1 | 0 | 0
  WBC, Missing | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Subjects With Normal or Abnormal Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: At Day 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
Participants
  ALT, Inside | 40 | 39 | 10 | 10 | 10
  ALT, Above | 0 | 1 | 0 | 0 | 0
  ALT, Below | 0 | 0 | 0 | 0 | 0
  ALT, Missing | 0 | 0 | 0 | 0 | 0
  AST, Inside | 40 | 39 | 10 | 10 | 10
  AST, Above | 0 | 1 | 0 | 0 | 0
  AST, Below | 0 | 0 | 0 | 0 | 0
  AST, Missing | 0 | 0 | 0 | 0 | 0
  Basophils, Inside | 40 | 40 | 10 | 10 | 10
  Basophils, Above | 0 | 0 | 0 | 0 | 0
  Basophils, Below | 0 | 0 | 0 | 0 | 0
  Basophils, Missing | 0 | 0 | 0 | 0 | 0
  Creatinine, Inside | 40 | 38 | 9 | 10 | 10
  Creatinine, Above | 0 | 1 | 0 | 0 | 0
  Creatinine, Below | 0 | 1 | 1 | 0 | 0
  Creatinine, Missing | 0 | 0 | 0 | 0 | 0
  Eosinophils, Inside | 38 | 38 | 10 | 10 | 10
  Eosinophils, Above | 2 | 2 | 0 | 0 | 0
  Eosinophils, Below | 0 | 0 | 0 | 0 | 0
  Eosinophils, Missing | 0 | 0 | 0 | 0 | 0
  Haemoglobin, Inside | 38 | 39 | 10 | 9 | 10
  Haemoglobin, Above | 0 | 0 | 0 | 0 | 0
  Haemoglobin, Below | 2 | 1 | 0 | 1 | 0
  Haemoglobin, Missing | 0 | 0 | 0 | 0 | 0
  Haematocrite, Inside | 38 | 40 | 10 | 10 | 10
  Haematocrite, Above | 0 | 0 | 0 | 0 | 0
  Haematocrite, Below | 2 | 0 | 0 | 0 | 0
  Haematocrite, Missing | 0 | 0 | 0 | 0 | 0
  Lymphocytes, Inside | 39 | 36 | 10 | 8 | 10
  Lymphocytes, Above | 1 | 2 | 0 | 1 | 0
  Lymphocytes, Below | 0 | 2 | 0 | 1 | 0
  Lymphocytes, Missing | 0 | 0 | 0 | 0 | 0
  Monocytes, Inside | 33 | 29 | 7 | 8 | 6
  Monocytes, Above | 7 | 11 | 3 | 2 | 4
  Monocytes, Below | 0 | 0 | 0 | 0 | 0
  Monocytes, Missing | 0 | 0 | 0 | 0 | 0
  Neutrophils, Inside | 39 | 39 | 10 | 9 | 10
  Neutrophils, Above | 0 | 0 | 0 | 0 | 0
  Neutrophils, Below | 1 | 1 | 0 | 1 | 0
  Neutrophils, Missing | 0 | 0 | 0 | 0 | 0
  Platelets, Inside | 38 | 38 | 10 | 9 | 10
  Platelets, Above | 0 | 0 | 0 | 0 | 0
  Platelets, Below | 2 | 2 | 0 | 1 | 0
  Platelets, Missing | 0 | 0 | 0 | 0 | 0
  RBC, Inside | 39 | 40 | 10 | 10 | 10
  RBC, Above | 0 | 0 | 0 | 0 | 0
  RBC, Below | 1 | 0 | 0 | 0 | 0
  RBC, Missing | 0 | 0 | 0 | 0 | 0
  WBC, Inside | 38 | 37 | 10 | 9 | 9
  WBC, Above | 0 | 0 | 0 | 0 | 0
  WBC, Below | 2 | 3 | 0 | 1 | 1
  WBC, Missing | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Subjects With Normal or Abnormal Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: At Day 37
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
Participants
  ALT, Inside | 39 | 39 | 10 | 10 | 10
  ALT, Above | 1 | 1 | 0 | 0 | 0
  ALT, Below | 0 | 0 | 0 | 0 | 0
  ALT, Missing | 0 | 0 | 0 | 0 | 0
  AST, Inside | 40 | 40 | 10 | 10 | 10
  AST, Above | 0 | 0 | 0 | 0 | 0
  AST, Below | 0 | 0 | 0 | 0 | 0
  AST, Missing | 0 | 0 | 0 | 0 | 0
  Basophils, Inside | 40 | 40 | 10 | 10 | 10
  Basophils, Above | 0 | 0 | 0 | 0 | 0
  Basophils, Below | 0 | 0 | 0 | 0 | 0
  Basophils, Missing | 0 | 0 | 0 | 0 | 0
  Creatinine, Inside | 39 | 38 | 10 | 10 | 10
  Creatinine, Above | 1 | 1 | 0 | 0 | 0
  Creatinine, Below | 0 | 1 | 0 | 0 | 0
  Creatinine, Missing | 0 | 0 | 0 | 0 | 0
  Eosinophils, Inside | 39 | 38 | 10 | 10 | 10
  Eosinophils, Above | 1 | 2 | 0 | 0 | 0
  Eosinophils, Below | 0 | 0 | 0 | 0 | 0
  Eosinophils, Missing | 0 | 0 | 0 | 0 | 0
  Haemoglobin, Inside | 38 | 39 | 10 | 9 | 10
  Haemoglobin, Above | 0 | 0 | 0 | 0 | 0
  Haemoglobin, Below | 2 | 1 | 0 | 1 | 0
  Haemoglobin, Missing | 0 | 0 | 0 | 0 | 0
  Haematocrite, Inside | 37 | 37 | 10 | 9 | 10
  Haematocrite, Above | 0 | 0 | 0 | 0 | 0
  Haematocrite, Below | 3 | 3 | 0 | 1 | 0
  Haematocrite, Missing | 0 | 0 | 0 | 0 | 0
  Lymphocytes, Inside | 38 | 38 | 10 | 10 | 9
  Lymphocytes, Above | 0 | 2 | 0 | 0 | 1
  Lymphocytes, Below | 2 | 0 | 0 | 0 | 0
  Lymphocytes, Missing | 0 | 0 | 0 | 0 | 0
  Monocytes, Inside | 30 | 35 | 9 | 7 | 7
  Monocytes, Above | 8 | 4 | 1 | 3 | 3
  Monocytes, Below | 2 | 1 | 0 | 0 | 0
  Monocytes, Missing | 0 | 0 | 0 | 0 | 0
  Neutrophils, Inside | 38 | 38 | 10 | 10 | 9
  Neutrophils, Above | 2 | 0 | 0 | 0 | 0
  Neutrophils, Below | 0 | 2 | 0 | 0 | 1
  Neutrophils, Missing | 0 | 0 | 0 | 0 | 0
  Platelets, Inside | 38 | 39 | 10 | 9 | 10
  Platelets, Above | 1 | 0 | 0 | 0 | 0
  Platelets, Below | 1 | 1 | 0 | 1 | 0
  Platelets, Missing | 0 | 0 | 0 | 0 | 0
  RBC, Inside | 40 | 40 | 10 | 10 | 10
  RBC, Above | 0 | 0 | 0 | 0 | 0
  RBC, Below | 0 | 0 | 0 | 0 | 0
  RBC, Missing | 0 | 0 | 0 | 0 | 0
  WBC, Inside | 37 | 39 | 10 | 9 | 10
  WBC, Above | 2 | 0 | 0 | 0 | 0
  WBC, Below | 1 | 1 | 0 | 1 | 0
  WBC, Missing | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Subjects With Normal or Abnormal Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: At Day 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
Participants
  ALT, Inside | 39 | 39 | 10 | 10 | 10
  ALT, Above | 0 | 1 | 0 | 0 | 0
  ALT, Below | 1 | 0 | 0 | 0 | 0
  ALT, Missing | 0 | 0 | 0 | 0 | 0
  AST, Inside | 38 | 40 | 10 | 10 | 9
  AST, Above | 2 | 0 | 0 | 0 | 1
  AST, Below | 0 | 0 | 0 | 0 | 0
  AST, Missing | 0 | 0 | 0 | 0 | 0
  Basophils, Inside | 40 | 40 | 10 | 10 | 10
  Basophils, Above | 0 | 0 | 0 | 0 | 0
  Basophils, Below | 0 | 0 | 0 | 0 | 0
  Basophils, Missing | 0 | 0 | 0 | 0 | 0
  Creatinine, Inside | 40 | 39 | 10 | 10 | 9
  Creatinine, Above | 0 | 0 | 0 | 0 | 0
  Creatinine, Below | 0 | 1 | 0 | 0 | 1
  Creatinine, Missing | 0 | 0 | 0 | 0 | 0
  Eosinophils, Inside | 38 | 38 | 10 | 10 | 10
  Eosinophils, Above | 2 | 2 | 0 | 0 | 0
  Eosinophils, Below | 0 | 0 | 0 | 0 | 0
  Eosinophils, Missing | 0 | 0 | 0 | 0 | 0
  Haemoglobin, Inside | 39 | 40 | 10 | 9 | 10
  Haemoglobin, Above | 0 | 0 | 0 | 0 | 0
  Haemoglobin, Below | 1 | 0 | 0 | 1 | 0
  Haemoglobin, Missing | 0 | 0 | 0 | 0 | 0
  Haematocrite, Inside | 38 | 36 | 10 | 9 | 10
  Haematocrite, Above | 0 | 0 | 0 | 0 | 0
  Haematocrite, Below | 2 | 4 | 0 | 1 | 0
  Haematocrite, Missing | 0 | 0 | 0 | 0 | 0
  Lymphocytes, Inside | 38 | 38 | 10 | 9 | 8
  Lymphocytes, Above | 2 | 0 | 0 | 0 | 1
  Lymphocytes, Below | 0 | 2 | 0 | 1 | 1
  Lymphocytes, Missing | 0 | 0 | 0 | 0 | 0
  Monocytes, Inside | 29 | 35 | 8 | 9 | 7
  Monocytes, Above | 11 | 5 | 2 | 1 | 3
  Monocytes, Below | 0 | 0 | 0 | 0 | 0
  Monocytes, Missing | 0 | 0 | 0 | 0 | 0
  Neutrophils, Inside | 39 | 36 | 10 | 10 | 8
  Neutrophils, Above | 0 | 2 | 0 | 0 | 1
  Neutrophils, Below | 1 | 2 | 0 | 0 | 1
  Neutrophils, Missing | 0 | 0 | 0 | 0 | 0
  Platelets, Inside | 39 | 38 | 10 | 10 | 10
  Platelets, Above | 0 | 0 | 0 | 0 | 0
  Platelets, Below | 1 | 2 | 0 | 0 | 0
  Platelets, Missing | 0 | 0 | 0 | 0 | 0
  RBC, Inside | 40 | 39 | 10 | 9 | 10
  RBC, Above | 0 | 0 | 0 | 1 | 0
  RBC, Below | 0 | 1 | 0 | 0 | 0
  RBC, Missing | 0 | 0 | 0 | 0 | 0
  WBC, Inside | 38 | 37 | 9 | 9 | 9
  WBC, Above | 0 | 1 | 0 | 0 | 0
  WBC, Below | 2 | 2 | 1 | 1 | 1
  WBC, Missing | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Levels of C-reactive Protein
Description: The levels of C-reactive protein are expressed in milligram per deciliter (mg/dL).
Time Frame: At Day 0
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
mg/dL | 0.10 [0.05 to 0.30] | 0.10 [0.10 to 0.30] | 0.15 [0.05 to 0.20] | 0.10 [0.05 to 0.10] | 0.30 [0.05 to 0.30]

14. Primary Outcome: Levels of C-reactive Protein
Description: The levels of C-reactive protein are expressed in milligram per deciliter (mg/dL).
Time Frame: At Day 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
mg/dL | 1.45 [0.65 to 2.35] | 1.05 [0.70 to 1.50] | 0.70 [0.60 to 1.00] | 0.10 [0.05 to 0.10] | 1.10 [0.60 to 1.70]

15. Primary Outcome: Levels of C-reactive Protein
Description: The levels of C-reactive protein are expressed in milligram per deciliter (mg/dL).
Time Frame: At Day 7
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
mg/dL | 0.20 [0.10 to 0.30] | 0.20 [0.10 to 0.30] | 0.20 [0.10 to 0.60] | 0.10 [0.05 to 0.20] | 0.15 [0.10 to 0.30]

16. Primary Outcome: Levels of C-reactive Protein
Description: The levels of C-reactive protein are expressed in milligram per deciliter (mg/dL).
Time Frame: At Day 30
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
mg/dL | 0.10 [0.05 to 0.20] | 0.10 [0.08 to 0.20] | 0.10 [0.05 to 0.20] | 0.10 [0.05 to 0.10] | 0.20 [0.10 to 0.40]

17. Primary Outcome: Levels of C-reactive Protein
Description: The levels of C-reactive protein are expressed in milligram per deciliter (mg/dL).
Time Frame: At Day 31
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
mg/dL | 1.65 [1.00 to 2.45] | 1.25 [0.80 to 2.05] | 1.15 [0.60 to 1.60] | 0.10 [0.05 to 0.20] | 0.75 [0.60 to 1.40]

18. Primary Outcome: Levels of C-reactive Protein
Description: The levels of C-reactive protein are expressed in milligram per deciliter (mg/dL).
Time Frame: At Day 37
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
mg/dL | 0.30 [0.20 to 0.60] | 0.20 [0.20 to 0.40] | 0.20 [0.20 to 0.30] | 0.10 [0.05 to 0.10] | 0.25 [0.10 to 0.40]

19. Primary Outcome: Levels of Immunoglobulin E
Description: The levels of Immunoglobulin E are expressed in 1000 units per liter (1000 U/L).
Time Frame: At Day 0
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: 1000 U/L
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
1000 U/L | 30.10 [14.85 to 160.50] | 61.55 [25.00 to 122.50] | 46.75 [14.90 to 99.80] | 39.55 [14.30 to 49.90] | 45.25 [28.20 to 82.40]

20. Primary Outcome: Levels of Immunoglobulin E
Description: The levels of Immunoglobulin E are expressed in 1000 units per liter (1000 U/L).
Time Frame: At Day 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: 1000 U/L
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
1000 U/L | 29.55 [13.80 to 159.00] | 61.90 [27.70 to 132.00] | 46.50 [13.60 to 95.30] | 41.05 [11.20 to 49.30] | 41.75 [30.10 to 78.80]

21. Primary Outcome: Levels of Immunoglobulin E
Description: The levels of Immunoglobulin E are expressed in 1000 units per liter (1000 U/L).
Time Frame: At Day 7
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: 1000 U/L
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
1000 U/L | 36.10 [14.60 to 160.50] | 65.50 [29.80 to 127.00] | 43.25 [13.80 to 78.50] | 38.00 [15.70 to 47.10] | 45.80 [27.70 to 77.60]

22. Primary Outcome: Levels of Immunoglobulin E
Description: The levels of Immunoglobulin E are expressed in 1000 units per liter (1000 U/L).
Time Frame: At Day 30
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: 1000 U/L
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
1000 U/L | 31.05 [13.70 to 149.00] | 58.60 [29.25 to 131.00] | 43.70 [15.90 to 66.90] | 38.10 [12.60 to 44.20] | 43.55 [27.10 to 67.90]

23. Primary Outcome: Levels of Immunoglobulin E
Description: The levels of Immunoglobulin E are expressed in 1000 units per liter (1000 U/L).
Time Frame: At Day 31
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: 1000 U/L
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
1000 U/L | 34.20 [14.90 to 156.00] | 64.10 [29.80 to 126.00] | 46.40 [14.40 to 71.20] | 39.05 [13.00 to 45.30] | 45.35 [25.70 to 72.30]

24. Primary Outcome: Levels of Immunoglobulin E
Description: The levels of Immunoglobulin E are expressed in 1000 units per liter (1000 U/L).
Time Frame: At Day 37
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: 1000 U/L
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
1000 U/L | 35.00 [14.30 to 159.50] | 60.35 [28.80 to 154.50] | 49.15 [16.40 to 77.10] | 40.85 [13.60 to 44.90] | 44.20 [26.10 to 68.80]

25. Secondary Outcome: Antibody Concentrations Against Mycobacterium Tuberculosis (M. Tuberculosis) Fusion Proteins M72 and Mtb72F
Description: Antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in Enzyme-Linked Immunosorbent Assay (ELISA) units per milliliter (EU/mL). The reference seropositivity cut-off values for anti-M72 and anti-Mtb72F antibodies were ≥ 2.8 EU/mL and ≥ 1.0 EU/mL, respectively.
Time Frame: At Day 0, prior to Dose 2 (Month 1), 1 month post-Dose 2 (Month 2) and Year 1 (Month 12)
Population: The analysis was performed on the According to protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
EU/mL
  Anti-M72, Day 0 | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4]
  Anti-M72, Month 1 | 24.7 [18.6 to 33.0] | 10.4 [7.8 to 13.8] | 14.4 [8.2 to 25.1] | 1.8 [1.0 to 3.0] | 1.4 [1.4 to 1.4]
  Anti-M72, Month 2: number analyzed (Participants) | 40 | 39 | 10 | 10 | 10
  Anti-M72, Month 2 | 722.6 [583.5 to 894.9] | 470.8 [394.0 to 562.5] | 491.9 [306.4 to 789.5] | 5.3 [1.5 to 18.2] | 1.4 [1.4 to 1.4]
  Anti-M72, Month 12 | 59.5 [48.8 to 72.6] | 42.5 [34.2 to 52.6] | 43.2 [25.3 to 73.8] | 2.7 [1.3 to 5.7] | 1.4 [1.4 to 1.4]
  Anti-Mtb72F, Day 0 | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 0.5]
  Anti-Mtb72F, Month 1 | 27.6 [20.8 to 36.8] | 11.5 [8.7 to 15.1] | 16.0 [9.3 to 27.8] | 0.8 [0.4 to 1.9] | 0.5 [0.5 to 0.5]
  Anti-Mtb72F, Month 12: number analyzed (Participants) | 40 | 39 | 10 | 10 | 10
  Anti-Mtb72F, Month 12 | 731.6 [589.0 to 908.8] | 473.1 [398.0 to 562.4] | 512.1 [314.6 to 833.6] | 3.2 [0.7 to 15.5] | 0.5 [0.5 to 0.5]
  Anti-Mtb72F, Month 2 | 44.7 [36.2 to 55.2] | 30.1 [24.4 to 37.1] | 31.6 [19.3 to 51.7] | 1.4 [0.5 to 3.8] | 0.5 [0.5 to 0.5]

26. Secondary Outcome: Antibody Concentrations Against M. Tuberculosis Fusion Protein M72
Description: Antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per milliliter (EU/mL). The reference seropositivity cut-off value for anti-M72 antibodies was ≥ 2.8 EU/mL.
Time Frame: At Year 2 (Month 24) and Year 3 (Month 36)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available at the Month 24 and Month 36 time points (M72/AS01B group and M72/AS02A group).
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | M72/AS01B Group | M72/AS02A Group
Number analyzed (Participants) | 31 | 37
EU/mL
  Anti-M72, Month 24 | 38.9 [29.5 to 51.1] | 21.6 [17.0 to 27.6]
  Anti-M72, Month 36: number analyzed (Participants) | 24 | 29
  Anti-M72, Month 36 | 29.2 [21.0 to 40.6] | 19.3 [14.0 to 26.6]

27. Secondary Outcome: Frequency of Mycobacterium Tuberculosis Fusion Protein (M72) Specific Cluster of Differentiation 4/8 (CD4/CD8+) T-cells Expressing at Least Two Different Cytokines
Description: Among cytokines expressed were interleukin-2 [IL-2] and/or interferon-gamma [IFN-γ] and/or tumour necrosis factor-alpha [TNF-α] and/or cluster of differentiation 40-ligand [CD40-L]. The analysis of cytokines expression was performed by flow cytometry using intracellular cytokine staining (ICS) on frozen peripheral blood mononuclear cell (PBMCs). Note: No vaccine induced responses were observed for CD8+ T-cells, so no results are presented throughout the record.
Time Frame: At Day 0, prior to Dose 2 (Month 1), 1 month post-Dose 2 (Month 2) and Year 1 (Month 12)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
CD4+ T-cells/million cells
  CD4+ All doubles, Day 0 | 90.5 [17.5 to 149.0] | 65.5 [1.0 to 121.5] | 58.0 [1.0 to 131.0] | 134.5 [1.0 to 186.0] | 45.0 [1.0 to 107.0]
  CD4+ All doubles, Month 1 | 955.5 [629.0 to 1395.0] | 484.0 [351.0 to 873.0] | 745.5 [515.0 to 818.0] | 173.0 [4.0 to 323.0] | 95.5 [30.0 to 160.0]
  CD4+ All doubles, Month 2: number analyzed (Participants) | 39 | 39 | 10 | 10 | 10
  CD4+ All doubles, Month 2 | 2641.0 [2029.0 to 4080.0] | 1589.0 [1206.0 to 2241.0] | 2082.5 [1451.0 to 2403.0] | 278.0 [80.0 to 514.0] | 43.0 [1.0 to 139.0]
  CD4+ All doubles, Month 12: number analyzed (Participants) | 39 | 39 | 9 | 10 | 10
  CD4+ All doubles, Month 12 | 1282.0 [940.0 to 1613.0] | 769.0 [492.0 to 1161.0] | 642.0 [504.0 to 758.0] | 153.5 [1.0 to 226.0] | 82.0 [1.0 to 165.0]

28. Secondary Outcome: Frequency of Mycobacterium Tuberculosis Fusion Protein (M72) Specific Cluster of Differentiation 4 (CD4+) T-cells Expressing at Least Two Different Cytokines
Description: Among cytokines expressed were interleukin-2 [IL-2] and/or interferon-gamma [IFN-γ] and/or tumour necrosis factor-alpha [TNF-α] and/or cluster of differentiation 40-ligand [CD40-L]. The analysis of cytokines expression was performed by flow cytometry using intracellular cytokine staining (ICS) on frozen peripheral blood mononuclear cell (PBMCs).
Time Frame: At Year 2 (Month 24) and Year 3 (Month 36)
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | M72/AS01B Group | M72/AS02A Group
Number analyzed (Participants) | 31 | 37
CD4+ T-cells/million cells
  CD4+ All doubles, Month 24 | 1506.0 [1000.0 to 2200.0] | 826.0 [520.0 to 1293.0]
  CD4+ All doubles, Month 36: number analyzed (Participants) | 24 | 26
  CD4+ All doubles, Month 36 | 1313.0 [1013.5 to 1886.5] | 507.0 [373.0 to 800.0]

29. Secondary Outcome: Frequency of M72 Specific CD4+ T-cells Expressing at Least One Cytokine and Another Signal Molecule
Description: Expressed cytokine combinations for CD4+ T-cells were CD40-L and interleukin-2 [IL-2] or interferon-gamma [IFN-γ] or tumour necrosis factor-alpha [TNF-α]; IL-2 and CD40-L, or IFN-γ, or TNF-α; IFN-γ and CD40-L, or IL-2, or TNF-α; TNF-α and CD40-L, or IL-2, or IFN-γ.
Time Frame: At Day 0, prior to Dose 2 (Month 1), 1 month post-Dose 2 (Month 2) and Year 1 (Month 12)
Population: as for outcome 27
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
CD4+ T-cells/million cells
  CD4+ CD40-L, Day 0 | 63.0 [27.5 to 146.5] | 50.0 [1.5 to 129.5] | 90.0 [1.0 to 156.0] | 81.5 [1.0 to 143.0] | 37.0 [1.0 to 89.0]
  CD4+ CD40-L, Month 1 | 883.0 [505.5 to 1282.0] | 420.5 [281.0 to 782.0] | 715.0 [435.0 to 818.0] | 158.5 [3.0 to 263.0] | 56.5 [28.0 to 137.0]
  CD4+ CD40-L, Month 2: number analyzed (Participants) | 39 | 39 | 10 | 10 | 10
  CD4+ CD40-L, Month 2 | 2333.0 [1877.0 to 3605.0] | 1466.0 [1077.0 to 2167.0] | 1997.5 [1413.0 to 2208.0] | 238.0 [102.0 to 418.0] | 29.0 [1.0 to 127.0]
  CD4+ CD40-L, Month 12: number analyzed (Participants) | 39 | 39 | 9 | 10 | 10
  CD4+ CD40-L, Month 12 | 1234.0 [881.0 to 1562.0] | 718.0 [474.0 to 1074.0] | 597.0 [496.0 to 694.0] | 137.0 [1.0 to 253.0] | 77.5 [1.0 to 166.0]
  CD4+ TNF-α, Day 0 | 65.0 [2.5 to 121.0] | 33.5 [1.0 to 79.5] | 45.0 [1.0 to 63.0] | 34.0 [1.0 to 204.0] | 40.5 [1.0 to 97.0]
  CD4+ TNF-α, Month 1 | 466.0 [330.0 to 684.5] | 250.0 [104.0 to 410.0] | 291.5 [243.0 to 465.0] | 59.0 [2.0 to 219.0] | 82.0 [35.0 to 113.0]
  CD4+ TNF-α, Month 2: number analyzed (Participants) | 39 | 39 | 10 | 10 | 10
  CD4+ TNF-α, Month 2 | 1394.0 [954.0 to 1964.0] | 744.0 [512.0 to 1293.0] | 863.0 [727.0 to 1133.0] | 110.5 [1.0 to 225.0] | 15.5 [1.0 to 111.0]
  CD4+ TNF-α, Month 12: number analyzed (Participants) | 39 | 39 | 9 | 10 | 10
  CD4+ TNF-α, Month 12 | 545.0 [377.0 to 821.0] | 321.0 [221.0 to 515.0] | 314.0 [166.0 to 434.0] | 50.0 [4.0 to 140.0] | 1.0 [1.0 to 76.0]
  CD4+ IL-2, Day 0 | 41.5 [2.0 to 107.5] | 44.5 [1.5 to 101.0] | 41.0 [1.0 to 156.0] | 50.5 [1.0 to 153.0] | 54.0 [1.0 to 74.0]
  CD4+ IL-2, Month 1 | 886.5 [494.5 to 1359.0] | 451.5 [297.0 to 762.0] | 732.0 [446.0 to 831.0] | 141.0 [1.0 to 254.0] | 62.0 [16.0 to 80.0]
  CD4+ IL-2, Month 2: number analyzed (Participants) | 39 | 39 | 10 | 10 | 10
  CD4+ IL-2, Month 2 | 2325.0 [1809.0 to 3338.0] | 1489.0 [1096.0 to 2107.0] | 1729.5 [1304.0 to 2130.0] | 223.5 [95.0 to 450.0] | 29.0 [1.0 to 138.0]
  CD4+ IL-2, Month 12: number analyzed (Participants) | 39 | 39 | 9 | 10 | 10
  CD4+ IL-2, Month 12 | 1212.0 [803.0 to 1530.0] | 650.0 [437.0 to 1054.0] | 569.0 [443.0 to 672.0] | 98.0 [1.0 to 212.0] | 77.5 [14.0 to 110.0]
  CD4+ IFN-γ, Day 0 | 34.5 [1.0 to 94.5] | 34.5 [1.0 to 70.0] | 35.0 [21.0 to 100.0] | 46.5 [1.0 to 75.0] | 57.0 [22.0 to 82.0]
  CD4+ IFN-γ, Month 1 | 168.5 [91.5 to 479.5] | 112.0 [41.0 to 197.0] | 107.0 [97.0 to 188.0] | 33.0 [1.0 to 138.0] | 62.5 [22.0 to 80.0]
  CD4+ IFN-γ, Month 2: number analyzed (Participants) | 39 | 39 | 10 | 10 | 10
  CD4+ IFN-γ, Month 2 | 820.0 [370.0 to 1277.0] | 275.0 [84.0 to 502.0] | 335.0 [148.0 to 529.0] | 58.0 [42.0 to 109.0] | 1.0 [1.0 to 33.0]
  CD4+ IFN-γ, Month 12: number analyzed (Participants) | 39 | 39 | 9 | 10 | 10
  CD4+ IFN-γ, Month 12 | 317.0 [164.0 to 471.0] | 109.0 [57.0 to 160.0] | 120.0 [59.0 to 224.0] | 27.5 [1.0 to 88.0] | 41.5 [1.0 to 72.0]

30. Secondary Outcome: Frequency of M72 Specific CD4+ T-cells Expressing at Least One Cytokine and Another Signal Molecule
Description: Expressed cytokine combinations for CD4+ T cells were CD40-L and interleukin-2 [IL-2] or interferon-gamma [IFN-γ] or tumour necrosis factor-alpha [TNF-α]; IL-2 and CD40-L, or IFN-γ, or TNF-α; IFN-γ and CD40-L, or IL-2, or TNF-α; TNF-α and CD40-L, or IL-2, or IFN-γ.
Time Frame: At Year 2 (Month 24) and Year 3 (Month 36)
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | M72/AS01B Group | M72/AS02A Group
Number analyzed (Participants) | 31 | 37
CD4+ T-cells/million cells
  CD4+ CD40-L, Month 24 | 1467.0 [973.0 to 1920.0] | 800.0 [520.0 to 1293.0]
  CD4+ CD40-L, Month 36: number analyzed (Participants) | 24 | 26
  CD4+ CD40-L, Month 36 | 1106.5 [900.0 to 1846.5] | 493.5 [373.0 to 773.0]
  CD4+ TNF-α, Month 24 | 574.0 [426.0 to 1226.0] | 307.0 [227.0 to 560.0]
  CD4+ TNF-α, Month 36: number analyzed (Participants) | 24 | 26
  CD4+ TNF-α, Month 36 | 833.5 [593.5 to 1170.0] | 293.0 [214.0 to 454.0]
  CD4+ IL-2, Month 24 | 1320.0 [906.0 to 1800.0] | 787.0 [520.0 to 1174.0]
  CD4+ IL-2, Month 36: number analyzed (Participants) | 24 | 26
  CD4+ IL-2, Month 36 | 1087.0 [799.5 to 1727.0] | 479.5 [307.0 to 693.0]
  CD4+ IFN-γ, Month 24 | 387.0 [226.0 to 894.0] | 200.0 [134.0 to 254.0]
  CD4+ IFN-γ, Month 36: number analyzed (Participants) | 24 | 26
  CD4+ IFN-γ, Month 36 | 373.0 [152.5 to 700.0] | 106.5 [66.0 to 187.0]

31. Secondary Outcome: Number of Subjects With Response to M72-specific CD4+ T-cells Secreting at Least Two Different Cytokines/Activation Markers
Description: The cut-off value used for analysis of the frequency of cells expressing cytokines/immune markers was the 313 CD4+ T-cells per million CD4+ T-cells, i.e. the 95th percentile of the pre-vaccination level of cells expressing cytokines/immune markers.
Time Frame: At Day 0, prior to Dose 2 (Month 1), 1 month post-Dose 2 (Month 2) and Year 1 (Month 12)
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
Participants
  Day 0 | 3 | 2 | 0 | 0 | 1
  Month 1 | 38 | 33 | 9 | 3 | 0
  Month 2: number analyzed (Participants) | 39 | 39 | 10 | 10 | 10
  Month 2 | 39 | 39 | 10 | 5 | 0
  Month 12: number analyzed (Participants) | 39 | 39 | 9 | 10 | 10
  Month 12 | 39 | 35 | 8 | 2 | 1

32. Secondary Outcome: Number of Subjects With Response to M72-specific CD4+ T-cells Secreting at Least Two Different Cytokines/Activation Markers
Description: as for outcome 31
Time Frame: At Year 2 (Month 24) and Year 3 (Month 36)
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01B Group | M72/AS02A Group
Number analyzed (Participants) | 31 | 37
Participants
  Month 24 | 31 | 36
  Month 36: number analyzed (Participants) | 24 | 26
  Month 36 | 24 | 23

33. Secondary Outcome: Concentrations of IFN-γ Produced in Serum Samples
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in picogram per milliliter (pg/mL). The reference seropositivity cut-off value was equal to or above (≥) 1 pg/mL.
Time Frame: Prior to (Day 0 and Day 30) and one day (Day 1 and Day 31) after each vaccination
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
Number analyzed (Participants) | 40 | 40 | 10 | 10 | 10
pg/mL
  IFN-γ, Day 0 | 0.6 [0.5 to 0.6] | 0.6 [0.5 to 0.6] | 0.6 [0.4 to 0.9] | 1.0 [0.4 to 2.2] | 1.0 [0.4 to 2.7]
  IFN-γ, Day 1 | 4.5 [2.8 to 7.1] | 1.0 [0.7 to 1.5] | 2.2 [0.7 to 6.6] | 0.7 [0.3 to 1.3] | 3.3 [0.8 to 14.2]
  IFN-γ, Day 30 | 0.6 [0.5 to 0.7] | 0.6 [0.5 to 0.7] | 0.6 [0.4 to 1.0] | 1.1 [0.4 to 2.7] | 1.1 [0.3 to 3.5]
  IFN-γ, Day 31: number analyzed (Participants) | 39 | 39 | 10 | 10 | 10
  IFN-γ, Day 31 | 77.2 [57.8 to 103.0] | 20.1 [13.2 to 30.4] | 23.4 [7.4 to 73.6] | 1.4 [0.5 to 3.8] | 4.1 [1.2 to 14.7]

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: during the 30-day (Days 0-29) post-vaccination period; SAEs: during the entire study period (from Day 0 up to Month 36) for the M72/AS01B Group and M72/AS02A Group, up to Month 12 for the Mtb72F/AS02A Group, Non-adjuvanted Group, and Control Group.
Arm/Group | M72/AS01B Group | M72/AS02A Group | Mtb72F/AS02A Group | Non-adjuvanted Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/40 | 0/40 | 1/10 | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 40/40 | 40/40 | 10/10 | 9/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M72/AS01B Group (N=40) | M72/AS02A Group (N=40) | Mtb72F/AS02A Group (N=10) | Non-adjuvanted Group (N=10) | Control Group (N=10)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M72/AS01B Group (N=40) | M72/AS02A Group (N=40) | Mtb72F/AS02A Group (N=10) | Non-adjuvanted Group (N=10) | Control Group (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 13 (15) | 4 (4) | 1 (1) | 2 (2) | 2 (2)
Fatigue (General disorders) | 36 (61) | 29 (46) | 8 (13) | 3 (4) | 6 (10)
Feeling of body temperature change (General disorders) | 2 (3) | 4 (6) | 1 (1) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 23 (27) | 10 (17) | 5 (6) | 2 (4) | 2 (3)
Genital candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 34 (61) | 27 (39) | 9 (17) | 4 (6) | 6 (13)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (9) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 10 (11) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site movement impairment (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site paraesthesia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 9 (9) | 4 (4) | 2 (4) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 3 (4) | 2 (2) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (12) | 8 (8) | 3 (3) | 3 (3) | 6 (6)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (6) | 1 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 40 (77) | 40 (77) | 10 (18) | 2 (3) | 10 (20)
Pyrexia (General disorders) | 25 (29) | 10 (12) | 4 (5) | 0 (0) | 1 (3)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Swelling (General disorders) | 9 (11) | 10 (17) | 5 (6) | 1 (1) | 3 (4)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.